CLINICAL TRIAL: NCT02291185
Title: Prediction of Fluid Responsiveness Using Dynamic Preload Indices During Arthroscopic Shoulder Surgery in the Beach Chair Position
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0698
Record Dates: First submitted 2014-10-30; First posted 2014-11-14 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Shoulder Arthroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The beach chair position (BCP) has been commonly used for shoulder arthroscopic surgery. Hemodynamic instability is frequently encountered problem associated with BCP. In addition, high rates of cerebral desaturation events have been reported during surgery in BCP. Although fluid loading could alleviate hypotension associated with BCP, it may lead to volume overload. As an alternative to static indices, dynamic preload indices such as pulse pressure variation (PPV) and stroke volume variation (SVV) were reported to be sensitive predictors of fluid responsivness in several surgical condition. The investigators will examine the abilities of PPV and SVV to predict fluid responsivness during shoulder arthroscopic surgery in BCP. Using transesophageal echocardiography (TEE), the investigators will directly estimate the change of cardiac output during BCP.

ELIGIBILITY:
Inclusion Criteria:

1. Above 20 years of age.
2. American Society of Anesthesiologists (ASA) Physical Status I, II, III.
3. shoulder arthroscopy under Beach-chair position

Exclusion Criteria:

1. severe functional liver or kidney disease
2. diagnosed HF ( NYHA class >3)
3. cerebrovascular disease 4. Pregnancy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing shoulder arthroscopic surgery in the beach chair position
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The changes between dynamic preload indices (SVV and PPV) and stroke volume index during beach chair position. We will measure them to evaluate the effect of beach chair position on PPV and SVV. | The participants will be followed up to 5 minutes after fluid challenge.
  To investigate the ability of SVV adn PPV to predict fluid responsiveness during beach chair position, using ROC curve.